CLINICAL TRIAL: NCT03739892
Title: Biomarkers to Predict Gain From Therapy in Motor Stroke
Acronym: GAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: C17-54
Record Dates: First submitted 2018-11-05; First posted 2018-11-14 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-03

CONDITIONS: Stroke; Motor Activity; Biomarker
MeSH Terms: conditions — Stroke; Motor Activity

STUDY DESIGN:
Intervention Model Description: physiopathological study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- stroke patients (Other): stroke patients with upper limb motor deficit receiving standard care of rehab
  Interventions: Behavioral: standard stroke rehabilitation

INTERVENTIONS:
Behavioral: standard stroke rehabilitation — standard rehabilitation according to the french standard care and to the severity of the patient

SUMMARY:
The aim is to determine predictors of treatment response, i.e gain from rehabilitation training, in post stroke upper limb deficits. The investigators will like to answer the following question: "What is this patient's potential for recovery, given his profile?" The investigators propose to conduct a longitudinal physiopathological study on the stroke patients with motor deficits who entered the rehab center of Pitié Salpêtrière hospital. The investigators will benefit from the organization, which is already in place (clinical asssessments and training) to add MRI, TMS and EEG recordings, as well as genotype analysis before the training offered in the rehabilitation unit. The investigators will repeat these assessments after the training (immeadiately and 6 weeks after).

DETAILED DESCRIPTION:
The protocol is based on 10 visits. The three main one are V1, V9 and V10. V1, V9 and V10 are the assessments visits with clinical scores, MRI TMS and EEG recordings. These are made before the training (V1), immediately after the 6 weeks of training (V9) and 6 weeks after (V10) V5 is a visit where the investigators will clinically assess the patients at three weeks of the training.

The other visits (V2, V3, V4, V6, V7, V8) consist in recording an EEG while patients are under training each week during six weeks.

ELIGIBILITY:
Inclusion Criteria:

(i) First-ever stroke patients (ii) Upper limb motor impairment (Fugl Meyer scale) (iii) post stroke delay between 7 and 42 days (iv) affiliated to french health care (v) Suitable for task based oriented training in the rehab center

Exclusion Criteria:

(i) age < 18 or > 85 years (ii) Hemianopia (iii) contra-indications to MRI or TMS assessments (iv) life threatening conditions (v) patients under legal protection (vi) pregnancy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2021-06-26 (Actual); Study Completion 2021-06-26 (Actual)

PRIMARY OUTCOMES:
Changes in a composite motor score post-pre training is the gain from therapy Candidates biomarkers: MRI, EEG, TMS, genotype | 6 weeks between pre and post assessment
  Changes in motor score Candidates biomarkers: MRI, EEG, TMS, genotypes post-pre training is the gain from therapy

SECONDARY OUTCOMES:
Changes in a composite motor score post-pre training is the gain from therapy | 12 weeks between pre and post assessment
  Changes in motor score Candidates biomarkers: MRI, EEG, TMS, genotypes post-pre training is the gain from therapy

CONTACTS AND LOCATIONS:
Locations (1):
- ICM, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jacquemont T, Valabregue R, Daghsen L, Moulton E, Zavanone C, Lamy JC, Rosso C. Association between superior longitudinal fasciculus, motor recovery, and motor outcome after stroke: a cohort study. Front Neurol. 2023 Jul 14;14:1157625. doi: 10.3389/fneur.2023.1157625. eCollection 2023. PMID 37521287